CLINICAL TRIAL: NCT00923065
Title: Data Collection, Clinical Care and Interventions in CCR, NCI
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040165; 04-C-0165; NCT00898625 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01-02

CONDITIONS: Neoplasms; Cancer
Keywords: Cancer; Natural History
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Consults: Individuals being seen as a consult.
- Donors: Donors of cellular products.
- Genetic Follow-Up: Individuals with a known/suspected germline genomic research incidental pathogenic or likely pathogenic variant, and/or who require CLIA confirmation.
- Patients: Individuals being enrolled for the treatment or follow-up of their disease.

SUMMARY:
This study provides cancer care through the National Cancer Institute's Medical Oncology Branch (MOB) to patients who are not enrolled in an active treatment research protocol. Patients receive standard treatments only; no investigational therapies are provided on this protocol.

Patients 18 years of age and older may be eligible for this protocol. Candidates are patients for whom an NCI investigator decides that the interests of the patient and the NCI are best served by the patient's enrollment in this protocol to receive care and follow-up within the MOB. This includes patients in the following categories:

* Patients previously enrolled in NCI trials whose participation in this protocol may continue to provide researchers important scientific information
* Patients who will be eligible for a research protocol within the foreseeable future
* Patients whose medical welfare will be seriously compromised by referral back to the community, such as patients with a rare or complex disease for which community resources are inadequate or unavailable
* Terminally ill patients who have received most of their specialized medical care at the Clinical Center and for whom humanitarian considerations dictate that they continue to receive their medical care at NIH after going off study for the remaining weeks or months of life
* Patients with cancer or HIV, or people at risk for cancer or HIV for whom cancer treatments at the NCI are requested through the MOB consult service
* Patients who are participating in a non-treatment NCI research protocol and require standard-of-care therapy
* Patients with cancer or HIV or people at risk for cancer for whom cancer treatment or management at the NCI would add significant value to the institute's cancer training program

Participants receive standard medical care, including periodic routine laboratory tests, diagnostic x-rays, and nuclear medicine scans to monitor the course of illness and the effects of any treatment.

DETAILED DESCRIPTION:
Background:

* Clinical Investigators within the Center for Cancer Research (CCR) at the National Cancer Institute (NCI) evaluate and treat patients with cancer, HIV, and individuals at risk for developing cancer in the context of active research protocols.
* In some cases, it may be in the best interests of both the individual and the CCR to provide consult services, treatment/interventions, and/or follow-up to certain individuals and collect the data obtained for future research.

Objectives:

-To provide a repository of information on enrolled participants to allow for hypothesis generation in future research

Eligibility:

* To allow a mechanism to provide consult, treatment, and medical follow-up for patients, including genetic education and counseling as well as cell/marrow donors to NCI patients and other individuals needed to be seen within the CCR.
* It is in the best interests of the individual and the CCR for the individual to receive a consultation or other medical evaluation, treatment, or follow-up, or to donate cellular products at the NCI, NIH Intramural Research Program.

Design:

* This protocol will provide the administrative vehicle for NCI investigators to provide consult services to individuals.
* Medical/surgical/radiotherapeutic care, treatment, and follow-up may be provided for certain participants.
* No investigational therapies will be administered on this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals must be age 2 years or older if therapeutic interventions are required. Otherwise, there are no age restrictions beyond the neonatal period (4 weeks).
* Individuals will be eligible if they meet one of the following criteria:

  * are seeking a consultation from NCI/CCR.
  * whose medical welfare will be seriously compromised by referral back to the community, such as rare/complex diseases in which community treatment is inadequate or adequate community resources are unavailable.
  * have cancer, HIV, or are at risk for cancer and/or HIV for whom cancer evaluation, treatment or management at the NCI is requested.
  * who will serve or have served as cellular therapy donors, for the treatment of a recipient of cellular therapy on an NCI trial.
  * are participants or biologic family members of deceased participants, where genetic testing is required or a clinically actionable germline pathogenic or likely pathogenic variant with medical implications was discovered by a research laboratory that requires CLIA confirmation. Note: In some cases, enrollment onto this study is also necessary when the prior study on which the involved participant was originally enrolled is closed and/or the participant is now off study.
* The individual or their Legally Authorized Representative is able and willing to provide informed consent.

EXCLUSION CRITERIA:

None

Ages: 4 Weeks to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals seen for appropriate clinical care evaluation and procedure, including: consultation, treatment and/or follow-up, cellular donation and/or genetic education, counseling, and CLIA confirmation of a germline research incidental pathogenic or likely pathogenic variant.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2004-06-10 (Actual)

PRIMARY OUTCOMES:
establishment of data repository for standard of care participants | ongoing
  Obtain and store information from participants seen for consult, treatment and medical follow-up for NCI patients, other Institute patients and individuals as specified.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima H Karzai, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-C-0165.html